CLINICAL TRIAL: NCT03688958
Title: Effect of Dietary Iodine Supplementation on the Proliferation of Breast Cancer
Brief Title: Iodine Supplementation on Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: Hospital General Regional #1 IMSS, Queretaro México (Unknown); Clínica Hospital Dr. Ismael Vázquez Ortiz ISSSTE, Queretaro Mexico (Unknown); Hospital Medico TEC100, Queretaro México (Unknown)
Responsible Party: Principal Investigator, Carmen Aceves, Investigador Titular, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INB-UNAM-004.H; IMSS-HGR1: 185-09-03-05/MPSS (Other: Hospital General Regional #1 IMSS); ISSSTE 22-205/CEI 248/2009 (Other: Clínica Hospital Dr. Ismael Vázquez Ortiz ISSSTE)
Record Dates: First submitted 2018-08-31; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Iodine

STUDY DESIGN:
Intervention Model Description: two randomized clinical groups including women with early (stage II) and advanced (stage III) breast cancer. In the Early group, women were treated with I2 (5 mg/day) or placebo (colored water) for 7 to 35 days. In the Advanced group, patients received treatment (I2 or placebo) along with 4 to 6 cycles of FEC/TE treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Early Cancer placebo (Placebo Comparator): The daily supplement of a vegetable colored water solution (drops) for 7 to 35 days in early breast cancer diagnosticated woman.
  Placebo: vegetable colored water solution (drops). Evaluate the activity of placebo on tumor size, and molecular tumor response, as well as side effects attenuation
  Interventions: Drug: Placebo
- Early Cancer Iodine (Experimental): The daily supplement of an iodine solution (drops, 5 mg/day) for 7 to 35 days in early breast cancer diagnosticated woman
  Interventions: Drug: iodine
- Advanced Cancer FEC/TE placebo (Placebo Comparator): The daily supplement of an vegetable colored water solution (drops) within 4 to 6 cycles of chemotherapy with FEC/TE in advanced breast cancer diagnosticated woman.
  Placebo: vegetable colored water solution (drops). Evaluate the adjuvancy of placebo in FEC/TE treatment on tumor size and molecular tumor response, as well as side effects attenuation.
  Interventions: Drug: FEC/TE Placebo
- Advanced Cancer FEC/TE + Iodine (Experimental): The daily supplement of an iodine solution (drops, 5 mg/day) within 4 to 6 cycles of chemotherapy with FEC/TE in advanced breast cancer diagnosticated woman Drug: Iodine solution (5 mg/day). Evaluate the adjuvancy of I2 on FEC/TE treatment on tumor size and molecular tumor response, as well as side effects attenuation.
  Other Name: evaluating the adjuvancy of iodine supplement in FEC/TE treatment
  Interventions: Drug: FEC/TE iodine

INTERVENTIONS:
Drug: Placebo — Selected patients with early breast cancer (stage II) non-pretreated received colored water solution (placebo) within the time before the hospital assigned them to her surgery (7 to 35 days).
  Other Names: control
  Arms: Early Cancer placebo
Drug: iodine — Selected patients with early breast cancer (stage II) non-pretreated received iodine solution (Experimental) within the time before the hospital assigned them to her surgery (7 to 35 days).
  Other Names: experimental
  Arms: Early Cancer Iodine
Drug: FEC/TE Placebo — The selected patients with advanced breast cancer (stage III) non-pretreated received colored water solution (placebo) within the time of oncology designed chemotherapy treatment FEC/TE (4 or 6 cycles/ every 21 days).
  Arms: Advanced Cancer FEC/TE placebo
Drug: FEC/TE iodine — The selected patients with advanced breast cancer (stage III) non-pretreated received iodine solution (experimental) within the time of oncology designed chemotherapy treatment (4 or 6 cycles/ every 21 days).
  Arms: Advanced Cancer FEC/TE + Iodine

SUMMARY:
The trial investigates the effect of oral supplement of molecular iodine (I2) alone and in combination with 4 to 6 cycles of FEC/TE (5-fluorouracil, epirubicin, cyclophosphamide/taxotere, epirubicin) treatment in woman diagnosticated with early (stage II) and advance (stage III) breast cancer, respectively. The study analyzes the clinical response [tumor size, thyroid status, side effects (Common Toxicity Criteria V4.0)] and molecular mechanisms in the tumor samples (transcriptomic, proteins and immune responses).

DETAILED DESCRIPTION:
The leading causes of failure of breast cancer treatment are the rapid development of metastases and tumor resistance to antineoplastic drugs. Anthracyclines (doxorubicin (DOX), epirubicin, etc.) are the golden standard in neoadjuvant therapy and are commonly used in the FEC/TE (5-fluorouracil, epirubicin, cyclophosphamide/taxotere, epirubicin) combination therapy during advanced breast cancer. However, even when treated with this potent chemotherapeutic combination, 30% of patients develop chemoresistance and cardiomyopathic side effects. Previous studies support that the oral supplement of molecular iodine (I2) exerts synergistic antineoplastic and cardioprotective impact when used in combination with the DOX in rodent and canine mammary cancer model. The present study performed two randomized clinical groups including women with early (stage II) and advanced (stage III) breast cancer. In the Early group, women were treated with I2 (5 mg/day) or placebo (colored water) for 7 to 35 days. In the Advanced group, patients received treatment (I2 or placebo) along with 4 to 6 cycles of FEC/TE treatment. The study analyzes the clinical response [tumor size, thyroid status, side effects (Common Toxicity Criteria V4.0)] and molecular mechanisms in the tumor samples (transcriptomic, proteins and immune responses).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, stage II or III breast cancer
* Scheduled to surgical of the primary tumor (stage II)
* Will receive neoadjuvant FEC/TE chemotherapy (stage III).
* age > 18 and < 81 years
* Non-pregnant
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Known sensitivity to iodine or FEC/TE
* Concurrent severe and/or uncontrolled disease
* Myocardial infarction within the last six months before the study
* Unstable or uncontrolled hypertension
* Thyroid dysfunction

Ages: 18 Years to 81 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-03-15 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Tumor response [change in size] | 20 minutes
  The size of the tumor is calculated by measuring the largest diameter of the tumor in the axial plane. The first measurement is obtained in the mammography taken before the start of the protocol and the second measurement is made on the tissue after surgery. The change percentage is obtained by dividing the final size between the initial size by 100.
Incidence of treatment-emergent adverse events [Safety and Tolerability]). | 40 minutes
  Presence or not of: Edema, hand-foot syndrome, anorexia, vomiting, diarrhea, nausea, asthenia (patient interview and clinical auscultation)
Differential Blood Count | 10 minutes (duration of blood withdrawal)]
  Differential blood count gives relative percentage of each type of white blood cell and helps reveal abnormal white blood cell populations (eg, blasts, immature granulocytes, or circulating mature cells in the peripheral blood).
Thyroid Test | 10 minutes (duration of blood withdrawal)
  Serum quantification of thyroxine, triiodothyronine, and thyroid stimulating hormone (nmol/ml) by ELISA Method
Cardiac damage | 10 minutes (duration of blood withdrawal)
  Measurement of creatine kinase myocardial band (CK-MB) concentration in serum (ImU/ml) by Colorimetric Method.
Iodine consumes | 10 minutes (duration of urine recollection)
  Measurement of iodine concentration in urine (ug/mL) by Ion Chromatography Method.
Tumor classification type and modification after treatment | 40 minutes
  Estrogen receptor (ER), Progesterone receptor (PR) and Human epidermal growth factor receptor 2 (HER2) presence in biopsy (initial) and tumor sample after treatments (final) by immunohistochemical method (number of positive cells/field).

SECONDARY OUTCOMES:
Disease-free survival | Every 6 months for 5 years
  The follow-up of the disease-free survival (DFS) at 5 years. (patient interview and clinical auscultation each six months)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Aceves, PhD, Principal Investigator — Universidad Nacional Autonoma de Mexico
Locations (3):
- Mexico (3):
  - Hospital Médico TEC100, Querétaro City, Querétaro
  - Clínica Hospital Dr. Ismael Vázquez Ortiz ISSSTE, Querétaro City, Querétaro
  - Hospital General Regional #1 IMSS, Querétaro City, Querétaro

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primarily and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Requestors will be required to sign a data access agreement

REFERENCES:
- [Result] Zambrano-Estrada X, Landaverde-Quiroz B, Duenas-Bocanegra AA, De Paz-Campos MA, Hernandez-Alberto G, Solorio-Perusquia B, Trejo-Mandujano M, Perez-Guerrero L, Delgado-Gonzalez E, Anguiano B, Aceves C. Molecular iodine/doxorubicin neoadjuvant treatment impair invasive capacity and attenuate side effect in canine mammary cancer. BMC Vet Res. 2018 Mar 12;14(1):87. doi: 10.1186/s12917-018-1411-6. PMID 29530037
- [Result] Bontempo A, Ugalde-Villanueva B, Delgado-Gonzalez E, Rodriguez AL, Aceves C. Molecular iodine impairs chemoresistance mechanisms, enhances doxorubicin retention and induces downregulation of the CD44+/CD24+ and E-cadherin+/vimentin+ subpopulations in MCF-7 cells resistant to low doses of doxorubicin. Oncol Rep. 2017 Nov;38(5):2867-2876. doi: 10.3892/or.2017.5934. Epub 2017 Sep 1. PMID 28901484
- [Result] Nava-Villalba M, Nunez-Anita RE, Bontempo A, Aceves C. Activation of peroxisome proliferator-activated receptor gamma is crucial for antitumoral effects of 6-iodolactone. Mol Cancer. 2015 Sep 17;14:168. doi: 10.1186/s12943-015-0436-8. PMID 26376791
- [Result] Alfaro Y, Delgado G, Carabez A, Anguiano B, Aceves C. Iodine and doxorubicin, a good combination for mammary cancer treatment: antineoplastic adjuvancy, chemoresistance inhibition, and cardioprotection. Mol Cancer. 2013 May 24;12:45. doi: 10.1186/1476-4598-12-45. PMID 23705792
- [Result] Aceves C, Anguiano B, Delgado G. The extrathyronine actions of iodine as antioxidant, apoptotic, and differentiation factor in various tissues. Thyroid. 2013 Aug;23(8):938-46. doi: 10.1089/thy.2012.0579. PMID 23607319
- [Result] Garcia-Solis P, Alfaro Y, Anguiano B, Delgado G, Guzman RC, Nandi S, Diaz-Munoz M, Vazquez-Martinez O, Aceves C. Inhibition of N-methyl-N-nitrosourea-induced mammary carcinogenesis by molecular iodine (I2) but not by iodide (I-) treatment Evidence that I2 prevents cancer promotion. Mol Cell Endocrinol. 2005 May 31;236(1-2):49-57. doi: 10.1016/j.mce.2005.03.001. Epub 2005 Apr 13. PMID 15922087

DOCUMENTS (1):
  • Informed Consent Form (2009-12-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT03688958/ICF_000.pdf